CLINICAL TRIAL: NCT03927066
Title: Physiological Validation of Current Machine Learning Models for Hemodynamic Instability in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Timothy B. Curry, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-002893
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Hypotension and Shock
MeSH Terms: conditions — Hypotension; Shock | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteer (Experimental): All Volunteers will be studied at rest and during experimental condition (lower body negative pressure)
  Interventions: Other: Assigned Interventions

INTERVENTIONS:
Other: Assigned Interventions — Simulated hypovolemia by applied suction to lower extremities to cause venous pooling.
  Other Names: Lower body negative pressure

SUMMARY:
This study will be collecting data on participants undergoing lower body negative pressure (LBNP) to simulate progressive blood loss. The goal of the study is to collect data to allow for development of an algorithm with machine learning to predict blood pressure responses to hyporvolemia by analyzing the arterial waveforms collected during LBNP.

DETAILED DESCRIPTION:
Death from exsanguination continues to be a major problem in combat casualty care and the care of civilians subjected to trauma. The ability to detect significant blood loss using traditional vital signs (heart rate, blood pressure) is marginal due to a variety of compensatory mechanisms that maintain blood pressure in the face of marked reductions in circulating blood volume. Along these lines, it is critical to develop monitoring devices and algorithms to non-invasively assess central blood volume in humans for the purposes of facilitating more timely interventions. The standard way to simulate hemorrhage in humans is to use Lower Body Negative Pressure (LBNP). In this technique, the lower body of a supine volunteer is enclosed in an airtight container while suction is applied to cause venous pooling in the legs and reduce central blood volume. This technique generates many physiological adaptations that are similar to that observed during blood loss studies in animals and human volunteers. Thus, the purpose of this study is to obtain data for use in developing monitoring technology to detect hemorrhage and other surrogate markers of central blood volume in humans.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese (BMI < 30)
* Non-smokers
* Free of any systemic diseases including hypertension, diabetes, coronary artery disease, neurologic disease, or any other major medical co-morbidity
* Women will be either surgically sterilized or non-pregnant as determined by a urine pregnancy test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | One day of study visit
  Arterial blood pressure both systolic and diastolic will be assessed prior to and during lower body negative pressure

SECONDARY OUTCOMES:
Heart rate | One day of study visit
  Heart rate prior to and during lower body negative pressure

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Curry, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials